CLINICAL TRIAL: NCT03160430
Title: A Two-Part Phase 2a Study in Patients With End-Stage Renal Disease Treated With Hemodialysis; Part A is an Open-Label Study Arm to Evaluate the Effect of Hemodialysis on the Pharmacokinetics of 100 mg RVX000222; and Part B is a Double-Blind, Randomized, Placebo-Controlled, Sequential Cross-Over Study Arm to Evaluate the Efficacy, Safety, and Pharmacokinetics of RVX000222
Brief Title: A Two-Part Phase 2a Study of RVX000222 in Patients With End-Stage Renal Disease Treated With Hemodialysis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVX222-CS-018
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Kidney Failure, Chronic
Keywords: Chronic Kidney Failure; ESRD; End-Stage Kidney Disease; End-Stage Renal Disease; Renal Disease, End-Stage; Renal Failure, Chronic; Renal Failure, End-Stage
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — apabetalone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A PK Arm (Experimental): a single 100 mg dose of RVX000222 (apabetalone) on the day of dialysis, followed by a one (1) week washout period, and a second dose of RVX000222 (apabetalone) administered on a non-dialysis day (total of two (2) 100 mg RVX000222 doses)
  Interventions: Drug: apabetalone
- Part B Sequence A (Placebo Comparator): RVX000222 (apabetalone) 100 mg b.i.d (total 200 mg/day) for 6 weeks; 4 Week Washout (No RVX000222/placebo administration); Placebo b.i.d for 6 weeks
  Interventions: Drug: apabetalone; Drug: Placebos
- Part B Sequence B (Placebo Comparator): Placebo b.i.d for 6 weeks; 4 Week Washout (No RVX000222/placebo administration); RVX000222 (apabetalone) 100 mg b.i.d (total 200 mg/day) for 6 weeks
  Interventions: Drug: apabetalone; Drug: Placebos

INTERVENTIONS:
Drug: apabetalone — RVX000222 oral (apabetalone), 100 mg capsule
  Other Names: RVX000222; RVX-208
Drug: Placebos — matching placebo capsule
  Other Names: Matching placebo
  Arms: Part B Sequence A; Part B Sequence B

SUMMARY:
This is a multi-center, two-part study; Part A and Part B. Part A of the study is an open-label, single-dose pharmacokinetic (PK) evaluation of 100 mg RVX000222 on dialysis and non-dialysis days in eight (8) End Stage Renal Disease (ESRD) patients who receive hemodialysis as standard of care.

Part B of the study is a double-blind, placebo-controlled study in up to thirty six (36) ESRD patients receiving hemodialysis using a sequential cross-over design with RVX000222 at a daily oral dose of 100 mg b.i.d. (200 mg per day) or matching placebo in combination with SoC.

The primary objective of the study is to evaluate if treatment with RVX000222 in combination with standard of care (SoC) decreases plasma alkaline phosphatase in comparison to placebo and SoC.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 and ≤80 years of age.
2. Diagnosis of end-stage renal disease and receiving hemodialysis an average of three (3) times per week for at least ninety (90) days prior to Enrollment/Visit 2.
3. Clinically stable, in the judgment of the investigator.
4. Female subjects must meet one of the following:

   1. If of childbearing potential, must have a negative serum pregnancy test and be willing and able to use medically acceptable non-hormonal method of birth control (non-hormonal intrauterine device, condom, or diaphragm) or remain abstinent from Screen until Follow-up Visit, or
   2. Be of non-child-bearing potential: post-surgical sterilization (hysterectomy or a bilateral oophorectomy) or post-menopausal. Post-menopausal is defined as amenorrhea for ≥2 years at Screen/Visit 1.
5. In the view of the investigator, during the course of the trial, subject is expected to:

   1. remain on unchanged standard of care medication from 4 weeks prior to Enrollment/Visit 2.
   2. not require hospitalization for any condition other than routine hemodialysis.
6. Have given signed informed consent to participate in the study.

Exclusion Criteria:

1. Planned major surgery in the next 4 months, including renal transplant, from Enrollment/Visit 2.
2. Major surgery, in the judgement of the investigator, within 12 weeks before enrollment/Visit 2 (excluding vascular access surgery).
3. Hospitalization for congestive heart failure, myocardial infarction, deep vein thrombosis, stroke or transient ischemic attack or peripheral arterial disease within 6 months before Enrollment/Visit 2.
4. New York Heart Association (NYHA) Classification, Class III or IV Heart Failure at Screen/Visit 1.
5. Diastolic blood pressure >110 mm Hg or systolic blood pressure >180 mm Hg during screen.
6. Currently receiving antibiotic therapy for systemic infection.
7. In the judgement of the Investigator, evidence of active hepatitis. Hepatitis serology testing will be performed at Screen/Visit 1.
8. History of malignancy of any organ system, treated or untreated, within the past 2 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
9. Red blood cell (RBC) transfusions within 12 weeks before Enrollment/Visit 2.
10. Current or recent (within 12 months prior to Visit 1) treatment with immunosuppressants (e.g., cyclosporine).
11. Use of fibrates at any dose or niacin/nicotinic acid 250 mg or more within 30 days prior to Screen/Visit 1.
12. Diagnosis of systemic hematologic disease (e.g., sickle cell anemia, myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia).
13. Hemoglobin <9.5 g/dL at Screen/Visit 1.
14. Alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN) at Screen/Visit 1.
15. Bilirubin >1.0 x ULN at Screen/Visit 1.
16. Pregnant or breast-feeding women.
17. Any condition which, in the opinion of the investigator, may place the subject at higher risk from his/her participation in the study, or is likely to prevent the subject from complying with the requirements of the study or completing the study.
18. Treatment with an investigational agent or device within 30 days or 5 half-lives before Enrollment/Visit 2 or scheduled to receive an investigational agent other than those specified by this protocol during the course of this study.
19. History of noncompliance with medical regimens or unwillingness to comply with the study protocol.
20. In the judgement of the Investigator, any disorder that may impact the ability to give informed consent for participation in this study.
21. Any condition that, in the opinion of the investigator, would confound the evaluation and interpretation of efficacy and/or safety data.
22. Persons directly involved in the execution of this protocol.

    Exclusion Criteria, Part A Only:
23. Are unwilling to abstain from alcoholic beverages, caffeine or xanthine-containing products (e.g., tea, coffee, chocolate, cola), and use of nicotine products from 24 hours prior to Clinical Research Unit (CRU) admission to 48 hours post RVX000222 dose administration.

Exclusion Criteria, Part B Only:

23. Parathyroid hormone, intact (PTH, intact) <150 pg/mL or >800 pg/mL at Screen/Visit 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-22 (Estimated); Primary Completion 2026-11-22 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
Percent change in alkaline phosphatase (ALP) concentration (Part B) | Percent change is computed relative to the beginning of each period (6 weeks)
  The primary endpoint of the study is the comparison of the RVX000222 treatment period to the placebo period in the percent change in ALP concentration. Percent change is computed relative to the beginning of each period.
Single Dose Cmax of RVX000222 (apabetalone) and the Metabolites RVX000288 and RVX000404 | 48 hours
  Primary PK comparison between dialysis (test) and non-dialysis (reference) days for Cmax of RVX000222 and its two principal metabolites, RVX000288 and RVX000404
Single Dose AUC of RVX000222 (apabetalone) and the Metabolites RVX000288 and RVX000404 | 48 hours
  Primary PK comparison between dialysis (test) and non-dialysis (reference) days for AUC of RVX000222 and its two principal metabolites, RVX000288 and RVX000404

SECONDARY OUTCOMES:
Changes in high-sensitivity C-Reactive Protein (hsCRP) | 6 weeks
  Changes in hsCRP in dialysis patients at the end of the RVX000222 treatment period relative to the end of the placebo period
Changes in Interleukin-13 (IL-13) | 6 weeks
  Changes in IL-13 in dialysis patients at the end of the RVX000222 treatment period relative to the end of the placebo period
Changes in Interleukin-6 (IL-6) | 6 weeks
  Changes in IL-6 in dialysis patients at the end of the RVX000222 treatment period relative to the end of the placebo period
Changes in Interleukin-8 (IL-8) | 6 weeks
  Changes in IL-8 in dialysis patients at the end of the RVX000222 treatment period relative to the end of the placebo period
Changes in Monocyte Chemoattractant Protein-1 (MCP-1) | 6 weeks
  Changes in MCP-1 in dialysis patients at the end of the RVX000222 treatment period relative to the end of the placebo period
Change in key markers of vascular mineralization | 6 weeks
  Change in key markers of vascular mineralization i.e. RANKL and osteoprotegerin at the end of the RVX000222 treatment period relative to the end of the placebo period
Changes in ALP isoenzymes | 6 weeks
  Changes in ALP isoenzymes at the end of the RVX000222 treatment period relative to the end of the placebo period
Changes in Parathyroid hormone (PTH) | 6 weeks
  Changes in parathyroid hormone at the end of the RVX000222 treatment period relative to the end of the placebo period
Change in apolipoprotein A1 (apoA-I), HDL-C, LDL-C, apolipoprotein B (apoB), and triglycerides | 6 weeks
  Change in apoA-I, HDL-C, LDL-C, apoB, and triglycerides at the end of the RVX000222 treatment period relative to the end of the placebo period
Change in Analyzing Data, Recognizing Excellence and Optimizing Outcomes All-Cause Mortality Risk Score For Patients on Chronic Hemodialysis (ARO Score) | 6 weeks
  Change in ARO Score at the end of the RVX000222 treatment period relative to the end of the placebo period

IPD SHARING:
Plan to Share IPD: Undecided